CLINICAL TRIAL: NCT04259190
Title: Does a Values Rationale Increase Willingness to Tolerate Distress in Interoceptive Exposure: Examination of a One-Session Randomized Clinical Trial
Brief Title: A Comparison of Treatment Rationales on Willingness to Tolerate Distress in Interoceptive Exposure
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Halted due to COVID-19.
Sponsor: Gina Boullion (Other)
Responsible Party: Sponsor-Investigator, Gina Boullion, Doctoral Candidate, University of Mississippi, Oxford
Organization: University of Mississippi, Oxford (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20-024
Record Dates: First submitted 2020-01-31; First posted 2020-02-06 (Actual); Last update posted 2020-06-26 (Actual); Status verified 2020-06

CONDITIONS: Anxiety Sensitivity
Keywords: anxiety sensitivity; panic; interoceptive exposure; exposure therapy; values

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Values rationale (Experimental): Interoceptive exposure exercises will be introduced as a way to help participants engage in more that they value.
  Interventions: Behavioral: interoceptive exposure
- Standard rationale (Active Comparator): Interoceptive exposure exercises will be introduced as a way to help participants experience less discomfort.
  Interventions: Behavioral: interoceptive exposure

INTERVENTIONS:
Behavioral: interoceptive exposure — Repeated 60-second trials of voluntary hyperventilation, each followed by a 15-second rest period. Participants will complete a minimum of 8 trials and continue additional trials until ratings of their most feared predicted outcome fall less than or below 5% likelihood.

SUMMARY:
The purpose of the current study is to examine the effect of emphasizing values in the treatment rationale on treatment response, willingness to tolerate distress, and acceptability of a one-session interoceptive exposure intervention for the reduction of anxiety sensitivity. A standard treatment rationale without values emphasis will serve as a control.

DETAILED DESCRIPTION:
Cognitive behavioral models of panic disorder maintain that recurrent, unexpected panic attacks result from anxiety sensitivity, or the fear of anxiety-related physiological sensations (e.g., fear of increased heart rate) and catastrophic misinterpretations regarding the danger of those sensations (e.g., misinterpreting increased heart rate as an oncoming heart attack). From these models and subsequent clinical research, interoceptive exposure has emerged as the most efficacious component of cognitive behavioral therapy for panic disorder treatment and, as expected, an efficacious intervention for decreasing anxiety sensitivity. Nevertheless, small-to-moderate effect sizes, wide variability in response rates and dropout rates indicated that panic disorder treatments may benefit from modifications to improve upon retention, response rates, and symptom reduction.

Patient motivation and lack of engagement have been identified as factors to intervene upon. Numerous therapeutic techniques have been used to facilitate patient motivation in treatment; however, one specific direction that has gained increasing empirical interest is the inclusion of values identification. Values have been incorporated as a motivational component in empirically supported behavioral techniques and treatments, including Motivational Interviewing, Behavioral Activation Treatment for Depression packages, and Acceptance and Commitment Therapy. Evidence from randomized controlled trials have generally supported the inclusion of packages containing values components in facilitating exposure therapy, and preliminary evidence has specifically favored the inclusion of packages containing values components in exposure therapy in cognitive behavioral therapy for panic disorder. However, there is no research known by the author that examines the influence of values on motivation in interoceptive exposure. Therefore, research examining the effect of a values component in isolation motivation in and acceptability of interoceptive exposure exercises has the potential to further improve treatment efficacy reducing costs associated with panic disorder and the many other conditions treated by interoceptive exposure. Therefore, the purpose of the current study is to examine the effect of emphasizing values in the treatment rationale on treatment response, willingness to tolerate distress, and acceptability of a one-session interoceptive exposure intervention among a clinical analogue sample with elevated anxiety sensitivity.

ELIGIBILITY:
Inclusion Criteria:

* Score ≥ 23 on the Anxiety Sensitivity Index - 3 (ASI-3)

Exclusion Criteria:

* Seizures
* Hypertension
* Heart problems
* Current pregnancy
* Asthma
* Other health conditions exacerbated by intense exercise

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-06-01 (Estimated); Primary Completion 2022-08-30 (Estimated); Study Completion 2022-08-30 (Estimated)

PRIMARY OUTCOMES:
Willingness to tolerate distress | change from pre-intervention to immediately post-intervention
  Willingness to tolerate distress will be assessed by identifying the activity item on the Albany Panic and Phobia Questionnaire (APPQ) - Agoraphobia subscale to which the participant responded with the highest score indicating most fear. The participant will then be asked, "How willing would you be to do [most feared activity] next week?" Responses will range from 0% to 100%.

SECONDARY OUTCOMES:
Straw breathing BAT peak fear ratings | pre-intervention
  Participants will be asked to engage in hyperventilation via breathing through a cocktail straw for three consecutive minutes pre-intervention. Participants will be asked to rate their peak fear ranging from 0 ("no fear") to 100 ("extreme fear or panic") on a 100-point visual analog scale after each minute. A peak fear rating will be calculated by computing the average of the three ratings.
Overbreathing BAT peak fear ratings | immediately post-intervention
  Participants will be asked to engage in one last overbreathing task post-intervention to see how long they can overbreathe. After discontinuation, participants will be asked to report their current level of fear ranging from 0 ("no fear") to 100 ("extreme fear or panic") on a 100-point visual analog scale.
Between trial fear ratings | change from pre-intervention to immediately post-intervention
  After each voluntary hyperventilation trial, participants will be asked to provide ratings of their peak fear. Participants will be asked to rate their peak fear during the trial ranging from 0 ("no fear") to 100 ("extreme fear or panic") on a 100-point visual analog scale.
Anxiety Sensitivity Index - 3 (ASI-3) | change from pre-intervention to immediately post-intervention
  The ASI-3 is an 18-item self-report measure of the fear of physiological arousal-related sensations. Scores on the ASI-3 can range from 0 to 72, with higher scores reflecting greater fear of arousal-related symptoms.
Albany Panic and Phobia Questionnaire (APPQ) | change from pre-intervention to immediately post-intervention
  The APPQ is a 27-item self-report measure of the fear of activities often avoided by individuals with agoraphobia and social phobia, and activities that typically produce physical sensations. Scores on the APPQ can range from 0 to 216, with higher scores reflecting higher levels of fear.
Between trial tolerability ratings | change from pre-intervention to immediately post-intervention
  After each voluntary hyperventilation trial, participants will be asked to provide ratings of tolerability of physiological sensations. Participants will be asked to rate the extent they perceived themselves as able to tolerate the physiological sensations during hyperventilation from 0 ("unable to tolerate them at all") to 100 ("completely able to tolerate them") on a 100-point visual analog scale.
Treatment Acceptability Questionnaire | immediately post-intervention
  A three-item self-report questionnaire was administered to participants to assess acceptability of the treatment provided. Participants will rate treatment acceptability, likeability, and aversiveness from "not at all" to "extremely" on a five-point Likert scale. Scores on the Treatment Acceptability Questionnaire can range from 0 to 12, with higher scores reflecting greater acceptability.

CONTACTS AND LOCATIONS:
Overall Officials: Gina Boullion, M.S., Principal Investigator — University of Mississippi Medical Center
Locations (1):
- University of Mississippi, University, Mississippi, United States

IPD SHARING:
Plan to Share IPD: No